CLINICAL TRIAL: NCT03007758
Title: Prospective Randomized Control Trial of Open Versus Robotic REtrOmuscular Ventral Hernia Repair (ORREO Trial)
Brief Title: Open Versus Robotic Retromuscular Ventral Hernia Repair
Acronym: ORREO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00062464
Record Dates: First submitted 2016-12-15; First posted 2017-01-02 (Estimated); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Ventral Hernia
Keywords: Hernia repair; Robotic hernia repair; Open hernia repair; Incisional hernia
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- robotic ventral hernia repair (VHR) (Active Comparator): Robotic VHR
  Interventions: Procedure: robotic ventral hernia repair
- open ventral hernia repair (VHR) (Active Comparator): Open VHR
  Interventions: Procedure: open ventral hernia repair

INTERVENTIONS:
Procedure: open ventral hernia repair — An open retromuscular ventral hernia repair involves an incision through your abdominal wall, most often through a prior surgery scar. The contents of the hernia, which may include intestine or fatty tissue, are returned into the abdominal cavity. The posterior (inner-most) layer of the abdominal wall is separated from the muscle and closed, which closes the abdominal cavity. Mesh is then placed over that closed layer, which is outside of the abdominal cavity, but below the abdominal muscles. The anterior (outer-most) layer of the abdominal wall is then closed over the mesh, which closes the hernia.
  Arms: open ventral hernia repair (VHR)
Procedure: robotic ventral hernia repair — A robotic retromuscular ventral hernia repair involves a similar separation of the layers of the abdominal wall, similar mesh placement, and similar closure of the hernia defect. The surgical robot is a tool that allows your surgeon to place long, narrow instruments through small incisions in order to perform surgery from the inside of your abdomen. Rather than one longer incision in the middle of your abdomen, four to six small incisions, about 1 inch, are made along the outer part of your abdomen between the rib cage and hip.
  Arms: robotic ventral hernia repair (VHR)

SUMMARY:
The purpose of this study is to determine how the robotic retromuscular hernia repair compares to the open retromuscular hernia repair for large hernia defects in patients at higher risk of wound complications.

DETAILED DESCRIPTION:
All patients presenting to the Greenville Health System Hernia Center who meet the inclusion criteria will be considered for enrollment. Patients who qualify and agree to participate will be randomized 1:1 to robotic retromuscular ventral hernia repair or open retromuscular ventral hernia repair. Data to be collected includes the following: demographic information, medical characteristics, medications, medical and surgical history, operative details, hospital stay data, and patient-reported outcomes via a quality of life questionnaire. Post-operative follow-up will occur at 2 weeks, 6 weeks, 6 months, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ventral or incisional hernia measuring ≥ 7 cm and ≤ 15 cm.
* At least one of the following risk factors: Body Mass Index > 30, Chronic Obstructive Pulmonary Disease, Diabetes Mellitus, current smoker (within 1 month)

Exclusion Criteria:

* Current abdominal wall infection
* Presence of ileostomy, colostomy, or ileal conduit
* Center for Disease Control wound class 3 or 4
* Hernia defect < 7 cm or >15 cm
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-12; Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy A Warren, MD, Principal Investigator — Prisma Health-Upstate

IPD SHARING:
Plan to Share IPD: Yes
All patients will be entered prospectively into the Americas Hernia Society Quality Collaborative (AHSQC) database.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After screening, 101 patients were consented.
Pre-assignment Details: One patient withdrew from the study prior to surgery, leaving 100 patients randomized for inclusion. A total of 7 patients were randomized but never went through with surgery (5 randomized to open, 2 randomized to robotic repair).
Period: Overall Study
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Started | 50 | 51
Randomization | 50 | 50
Surgery | 48 | 45
Completed 30-Day Follow-up | 45 | 44
Analysis of 30-day Outcomes | 46 | 44
Analysis of 2-year Outcomes | 32 | 30
Completed | 32 | 30
Not Completed | 18 | 21

BASELINE CHARACTERISTICS:
Population: After screening, 101 patients were consented. One patient withdrew from the study prior to surgery, leaving 100 patients randomized for inclusion. A total of 7 patients were randomized but never went through with surgery (5 randomized to open, 2 randomized to robotic repair). Two patients in the robotic arm and one in the open arm did not complete 30-day follow-up and were excluded, leaving 46 rRMVHR and 44 RMVHR patients for analysis of the primary outcome.
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR) | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 14 | 12 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 18 | 14 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 42 | 43 | 85
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 37 | 40 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Comorbidities [Count of Participants; unit: Participants]
  HTN | 26 | 28 | 54
  DM | 13 | 16 | 29
  COPD | 7 | 6 | 13
Active Smoker [Count of Participants; unit: Participants] | 16 | 14 | 30
ASA [Count of Participants; unit: Participants] — ASA I: A person in good health. ASA II: A mild but well-managed or treated condition. ASA III: A serious condition that has an impact on a person's overall health. ASA IV: A severe condition that's life-threatening. ASA V: A life-threatening condition that needs immediate surgery to increase survival odds.
  ASA VI: A deceased person who is an organ donor.
  Participants
    2 | 13 | 12 | 25
    3 | 32 | 32 | 64
    4 | 1 | 0 | 1
Hernia Type [Count of Participants; unit: Participants] — Participants can be counted more than once in the incisional and recurrent hernia categories.
  Participants
    Incisional | 44 | 41 | 85
    Primary Ventral | 2 | 1 | 3
    Parastomal | 0 | 2 | 2
    Recurrent Hernia | 16 | 23 | 39
Number of Prior Repairs [Count of Participants; unit: Participants]
  None | 30 | 21 | 51
  1 | 10 | 20 | 30
  2 | 5 | 2 | 7
  3 or more | 1 | 1 | 2
Prior Mesh Present [Count of Participants; unit: Participants] | 7 | 16 | 23
Myofascial release [Count of Participants; unit: Participants] — 34 patients in the open arm received a posterior rectus sheath release only. 32 patients in the robotic arm received a posterior rectus sheath release only. 14 patients in the robotic arm and 10 patients in the open received a transversus abdominis release.
  Participants
    Posterior rectus sheath only | 32 | 34 | 66
    Transversus Abdominis Release | 14 | 10 | 24
Intraoperative Complications [Count of Participants; unit: Participants] | 6 | 4 | 10
Bowel Injury (serosa) [Count of Participants; unit: Participants] | 6 | 2 | 8
Bowel Injury (full-thickness) [Count of Participants; unit: Participants] | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Composite Outcome of Diagnosis of Surgical Site Occurrence or Infection, Hospital Readmission, or Hernia Recurrence
Description: A composite outcome of events which are clinically significant including but not limited to seroma requiring procedural intervention, skin dehiscence, cellulitis, hematoma, skin necrosis, and surgical site infections which may require interventions such as wound care or antibiotic therapy.
Time Frame: Through study completion, an average of 2 years
Population: After screening, 101 patients were consented. One patient withdrew from the study prior to surgery, leaving 100 patients randomized for inclusion. A total of 7 patients were randomized but never went through with surgery (5 randomized to open, 2 randomized to robotic repair). Two patients in the robotic arm and one in the open arm did not complete 30-day follow-up and were excluded, leaving 46 robotic RMVHR and 44 open RMVHR patients for analysis of the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
Participants | 9 | 9

2. Secondary Outcome: All Surgical Site Occurrences
Description: Surgical site occurrence (SSO) is defined as all wound complications that occur after a surgical procedure but are not surgical site infections.
Time Frame: Post-operatively: 2 weeks, 6 weeks, 6 months, 1 year, 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
Participants | 8 | 7

3. Secondary Outcome: Surgical Site Occurrences Requiring Procedural Intervention
Description: as for outcome 2
Time Frame: Post-operatively: 2 weeks, 6 weeks, 6 months, 1 year, 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
Participants | 6 | 3

4. Secondary Outcome: All Surgical Site Infections
Description: Surgical site occurrence is defined as all wound complications that occur after a surgical procedure but are not surgical site infections.
Time Frame: Post-operatively: 2 weeks, 6 weeks, 6 months, 1 year, 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
Participants | 2 | 3

5. Secondary Outcome: Surgical Site Infections Requiring Procedural Intervention
Time Frame: Post-operatively: 2 weeks, 6 weeks, 6 months, 1 year, 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
Participants | 6 | 3

6. Secondary Outcome: Length of Stay at Hospital Measured in Days
Time Frame: Time from procedure until discharge, an expected range of 2 to10 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
days | 1 [0 to 5] | 2 [0 to 5]

7. Secondary Outcome: Operative Time (Procedure Start to Procedure Finish Measured in Minutes)
Time Frame: Day of surgery
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
minutes | 206 [184 to 237] | 156 [130 to 205]

8. Secondary Outcome: Cost for Hospital Charges From Billing Office
Time Frame: Through study completion, an average of 2 years
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: U.S. Dollars
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
U.S. Dollars | 11747 [9717 to 13530] | 9267 [8873 to 11641]

9. Secondary Outcome: BMI
Description: Body Mass Index
Time Frame: Measured at study enrollment
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
kg/m^2 | 36.7 [30.6 to 41.9] | 36.7 [31.6 to 40.2]

10. Secondary Outcome: Hernia Width
Description: Width of Hernia
Time Frame: measured at surgery
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
cm | 8 [6 to 10] | 10 [8 to 12]

11. Secondary Outcome: Hernia Length
Description: Length of Hernia
Time Frame: measured at surgery
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 44
cm | 15 [12 to 20] | 15 [10 to 19]

12. Secondary Outcome: Quality of Life Via Questionnaire - 30 Days
Description: Patient reported outcomes via the Hernia related quality of life score. The survey contains 12 statements about the patients abdominal wall and asks the patient to rate how strongly the disagree (1) or agree (6) with the statements on a scale 1-6. The score is calculated with the following formula: (120-[(20/12)*(sum of response on all 12 questions)]).The highest possible number, meaning the abdominal wall does not affect the patient, is 100, and the lowest, meaning the abdominal wall greatly affects the patient's quality of life, is a 0.
Time Frame: assessed at Baseline and Post-operatively at 30 days
Population: 41 patients in the robotic arm completed the 30 day PROs and 41 patients in the open arm completed the 30 day PROs.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 41 | 41
units on a scale
  Baseline Patient Reported Outcomes | 34 [16 to 52] | 28 [16 to 64]
  30 Day Patient Reported Outcomes | 38 [18 to 68] | 50 [34 to 58]
  Difference | 0 [-22 to 32] | 16 [-20 to 30]

13. Secondary Outcome: Quality of Life Via Questionnaire - 6 Through 12 Months
Description: Patient reported outcomes via the Hernia related quality of life score. The survey contains 12 statements about the patients abdominal wall and asks the patient to rate how strongly the disagree (1) or agree (6) with the statements on a scale 1-6.The score is calculated with the following formula: (120-[(20/12)*(sum of response on all 12 questions)]).The highest possible number, meaning the abdominal wall does not affect the patient, is 100, and the lowest, meaning the abdominal wall greatly affects the patient's quality of life, is a 0.
Time Frame: assessed at Baseline and Post-operatively at 6 through 12 months. Data for the 6 and 12-month patient reported outcomes were combined for analysis.
Population: 39 patients in the robotic arm completed the 6 or 12 month PROs and 33 patients in the open arm completed the 6 or 12 month PROs. Data collected at both 6 month and 12 month time points but they were combined for analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 39 | 33
units on a scale
  Baseline Patient Reported Outcomes | 26 [12 to 40] | 46 [34 to 80]
  6-12 month Patient Reported Outcomes | 86 [64 to 94] | 90 [72 to 96]
  Difference | 60 [22 to 78] | 20 [10 to 54]

14. Secondary Outcome: Quality of Life Via Questionnaire - 24 Months
Description: Patient reported outcomes via the Hernia related quality of life score. The survey contains 12 statements about the patients abdominal wall and asks the patient to rate how strongly the disagree (1) or agree (6) with the statements on a scale 1-6. The score is calculated with the following formula: (120-[(20/12)*(sum of responses on all 12 questions)]).The highest possible number, meaning the abdominal wall does not affect the patient, is 100, and the lowest, meaning the abdominal wall greatly affects the patient's quality of life, is a 0.
Time Frame: assessed at Baseline and Post-operatively at 24 months
Population: 32 patients in the robotic arm completed the 24 month patient reported outcomes and 30 patients in the open arm completed the 24 month patient reported outcomes.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 32 | 30
units on a scale
  Baseline Patient Reported Outcomes | 36 [21 to 69] | 32 [16 to 50]
  24 month Patient Reported Outcomes | 80 [42 to 92] | 91 [76 to 94]
  Difference | 28 [-5 to 56] | 59 [14 to 64]

15. Secondary Outcome: Pain Score - 30 Day Patient Reported Outcomes
Description: Patient is asked 3 different questions all in relation to their pain in the past 7 days: how intense was it as its worst, on average, and right now. They then rank their pain for each question on a scale of 1 - 5. 1 meaning no pain and 5 very severe pain. The pain scores were then averaged and used for this analysis.
Time Frame: assessed at Baseline and Post-operatively at 30 days.
Population: 41 patients in the robotic arm completed the 24 month patient reported outcomes and 41 patients in the open arm completed the 24 month patient reported outcomes.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 41 | 41
units on a scale
  Baseline Patient Reported outcomes | 2 [1 to 2] | 3 [2 to 3]
  30 Day Patient reported outcomes | 3 [2 to 3] | 2 [2 to 3]
  Difference | 1 [0 to 2] | 0 [-1 to 1]

16. Secondary Outcome: Pain Score - 6 or 12 Month Patient Reported Outcomes
Description: as for outcome 15
Time Frame: assessed at Baseline and Post-operatively at 6-12 months; data for 6 and 12-month pain scores were combined for analysis.
Population: 39 patients in the robotic arm completed the 6 or 12 month patient reported outcomes and 33 patients in the open arm completed the 6 or 12 month patient reported outcomes. Data collected at both 6 month and 12 month time points but they were combined for analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 39 | 33
units on a scale
  Baseline Patient Reported outcomes | 2 [2 to 3] | 2 [1 to 3]
  6 or 12 month Patient reported outcomes | 1 [1 to 2] | 1 [1 to 2]
  Difference | -1 [-2 to 0] | -1 [-1 to 0]

17. Secondary Outcome: Pain Score - 24 Month Patient Reported Outcomes
Description: as for outcome 15
Time Frame: assessed at Baseline and Post-operatively at 24 months
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 32 | 30
units on a scale
  Baseline Patient Reported outcomes | 2 [2 to 3] | 2 [2 to 3]
  24 month Patient reported outcomes | 1 [1 to 2] | 1 [1 to 1]
  Difference | -1 [-1.5 to 0] | -1 [-2 to 0]

18. Secondary Outcome: Ventral Hernia Recurrence Inventory 1 Year
Description: Patients are asked 3 yes or no questions about their hernia operation: do you feel your hernia has come back, do you feel or see a bulge, and do you have physical pain or symptoms at the site.
Time Frame: assessed at Baseline and Post-operatively at 12 months.
Population: 39 patients in the robotic arm completed the 12 month patient reported outcomes and 33 patients in the open arm completed the 12 month patient reported outcomes.
Measure: Number; unit: count of "yes" answers
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 39 | 33
count of "yes" answers
  Pain at hernia site | 9 | 5
  Bulging at hernia site | 16 | 7
  Do you feel your hernia has come back? | 2 | 2

19. Secondary Outcome: Ventral Hernia Recurrence Inventory 2 Years
Description: as for outcome 18
Time Frame: assessed at Baseline and Post-operatively at 24 months
Population: as for outcome 14
Measure: Number; unit: count of "yes" answers
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 32 | 30
count of "yes" answers
  Pain at hernia site | 8 | 4
  Bulging at hernia site | 11 | 3
  Do you feel your hernia has come back? | 7 | 1

20. Secondary Outcome: Hernia Recurrence
Description: The ventral hernia recurrence inventory asked patients if they have had any additional surgery since the hernia operation. If they answer yes, they choose if the surgery was for a hernia or another reason. The answers from 1 year follow up and 2 year follow up to the last question were combined for this analysis. Composite recurrence was then determined by excluding patients with negative CT scan or physical exam but had answered the ventral hernia recurrence inventory indication the hernia recurrence.
Time Frame: assessed Post-operatively as 24 months
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 32 | 30
Participants
  Ventral Hernia Recurrence Inventory - Recurrence at 2 years | 11 | 4
  Composite Recurrence | 4 | 1

21. Secondary Outcome: Conversion to Open
Description: Robotic surgeries converted to open surgeries.
Time Frame: Assessed at index surgery.
Population: Patient who are randomized to receive an open ventral hernia repair were not assessed for Conversion to Open
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
Number analyzed (Participants) | 46 | 0
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow up (2 years after surgery)
Arm/Group | Robotic Ventral Hernia Repair (VHR) | Open Ventral Hernia Repair (VHR)
All-Cause Mortality (participants affected / at risk) | 2/50 | 2/51
Serious Adverse Events (participants affected / at risk) | 9/50 | 6/51
Other Adverse Events (participants affected / at risk) | 15/50 | 7/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Robotic Ventral Hernia Repair (VHR) (N=50) | Open Ventral Hernia Repair (VHR) (N=51)
Hematoma (Surgical and medical procedures) | 3 (3) | 0/50 (0) — Pt was admitted to the hospital on 5/3/2018 for dizziness, blurred vision, and weakness. A CT scan was performed which showed a large hematoma at abdominal wall. Pt was put on anticoagulant Eliquis and discharged on 5/5/2018.
small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) — bowel obstruction due to adhesions
Wound infection (Surgical and medical procedures) | 1 (1) | 3 (3) — wound infection that required inpatient care and drainage
Intraperietal hernia (Surgical and medical procedures) | 1 (1) | 0 (0) — Patient complained of a bursting, pulling sensation in her abdomen. CT scan showed an intraparietal hernia which was repaired
Post surgical spine infection (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient to orthopedic spine surgery service for the diagnosis of acute paraplegia secondary to post-surgical infection.
Motor vehicle accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient visited ER after MVC; fractured right acetabular and multiple rib fractures
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) — patient complaining of chest pain
Total left hip anthroplast (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — patient had hip replacement
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Ventral Hernia Repair (VHR) (N=50) | Open Ventral Hernia Repair (VHR) (N=51)
Seroma (Surgical and medical procedures) | 6 (6) | 0 (0) — Patient developed a seroma. Patient came back into office and provider aspirated the seroma. Patient came back into office for their final study visit and provider again aspirated the seroma
progressive renal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) — Pt had known history of kidney disease and required dialysis post-operatively
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Patient developed fibrillation during dialysis
Enterotomies (Surgical and medical procedures) | 0 (0) | 1 (1) — bowel enterotomies occurred during intraoperative lysis of adhesions
Hematoma (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient's incision began to drain.
inguinal hernia repair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — patient had groin pain and CT scan showed inguinal hernia. Repaired with surgery
Superficial skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Cellulitis near incision
Whiplash (Nervous system disorders) | 1 (1) | 0 (0) — whiplash due to MVA
Abdominal pain (Surgical and medical procedures) | 2 (2) | 1 (1) — reports abdominal pain or tenderness
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) — patient went to cardiology for chest pain and diagnosed with CAD
Ureteral stone (Renal and urinary disorders) | 0 (0) | 1 (1) — patient reported flank and abdominal pain. CT scan showed ureteral stone
abdominal wall bulge (Surgical and medical procedures) | 1 (1) | 0 (0) — patient reported abdominal wall bulge
rectal bleeding (Renal and urinary disorders) | 1 (1) | 0 (0) — blood in stool and rectal bleeding
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — patient reported constipation that lead to diarrhea and vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT03007758/Prot_SAP_000.pdf